CLINICAL TRIAL: NCT04370171
Title: Management of Diabetic Patients With Telemedicine in the Context of the Covid-19 Epidemic: Prospective Observational Study
Brief Title: Management of Diabetic Patients With Telemedicine in the Context of the Covid-19 Epidemic
Acronym: TeleCoviDiab
Status: Completed | Type: Observational
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Other Study IDs: 7775
Record Dates: First submitted 2020-04-27; First posted 2020-04-30 (Actual); Last update posted 2020-11-10 (Actual); Status verified 2020-04

CONDITIONS: Diabetes; Covid-19
Keywords: Diabetes; Telemedicine; Covid-19 epidemic; Glucose control
MeSH Terms: conditions — Diabetes Mellitus; COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Group TC: Diabetic patients followed by Teleconsultation: Teleconsultation group will be composed of patients for whom the consultation initially scheduled in the presence of the diabetologist has been replaced by a teleconsultation due to the availability of diabetologists whose activity is focused on the management of Covid-19 negative patients.
  Interventions: Other: Teleconsultation either by phone or by computer consultation
- Group P: Diabetic patients with conventional follow-up: Conventional group will be composed of patients for whom the consultation initially scheduled in the presence of the diabetologist was differed by 6 months due to the activity of some diabetologists entirely redirected towards the management of Covid-19 positive patients and not available
  Interventions: Other: care modalities

INTERVENTIONS:
Other: care modalities — For these patients the consultation has been postponed for 6 months. No specific intervention for this group of patient.
  Groups: Group P: Diabetic patients with conventional follow-up
Other: Teleconsultation either by phone or by computer consultation — Management of diabetic patients by telemedicine with a teleconsultation either by phone or by computer consultation
  Groups: Group TC: Diabetic patients followed by Teleconsultation

SUMMARY:
Since the end of February 2020, Covid-19 infection has spread widely in France, particularly in the East region, with on March 25th, 2020, 5,479 infected patients and 407 deceased patients, including 256 in Alsace. Among the hospitalized patients reported in the initial Chinese studies, 48% had co-morbidity, particularly diabetes or cardiovascular disease. Covid-19 infection does not appear to be more common in diabetic patients, but infected diabetics have more severe forms.

The prevalence of diabetes is high in Alsace affecting 6.5% of the population against 4.6% in France. Du to health containment measures, asymptomatic diabetic patients can no longer come to the clinic in Hospital for their consultation. However, in the current epidemiological context, maintaining optimal glycemic control is fundamental since some of diabetic patients will have Covid-19 infections. Furthermore, the sedentary lifestyle and snacking linked to the confinement period will contribute to a glycemic imbalance in some patients. Telemedicine, and in particular teleconsultation, which until now has been very uncommon in the management of diabetic patients, represents a very interesting alternative for monitoring these patients and maintaining satisfactory metabolic control during the current period of confinement and Covid-19 epidemic.

ELIGIBILITY:
Inclusion Criteria:

* Adult diabetic patient (type 1,2, MODY, secondary, post transplantation) followed by diabetology consultation at the hospital or by a liberal diabetologist
* Subject affiliated to a social health insurance
* Subject able to understand the objectives of the research
* Subject who expressed his non opposition to the research

Exclusion Criteria:

* Pregnant woman
* Patients with acute complications (foot ulcer, post stroke, post IDM)
* Cancer or life expectancy of less than 6 months
* Inability to provide informed information to the subject (subject in an emergency, difficulty of understanding for the subject, etc.)
* Subject under judicial protection
* Subject under guardianship or curatorship

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Diabetic patients regularly followed in a clinic at the University Hospital of Strasbourg or followed by a liberal diabetologist in Strasbourg
Sampling Method: Non-Probability Sample
Enrollment: 610 (Actual)
Dates: Start 2020-05-04 (Actual); Primary Completion 2020-05-29 (Actual); Study Completion 2020-05-29 (Actual)

PRIMARY OUTCOMES:
Comparison of metabolic control (HbA1C) between diabetic patients followed by teleconsultation and patients with a conventional follow-up during Covid-19 infection. | HbA1C measured at 3 months post-telemedicine consultation group / post-cancellation of the face-to-face consultation group (variation versus basal)
  In the Covid 19 epidemic context, the face-to-face consultation of diabetic patients with the hospital's physician or their diabetologist is / will be replaced by a teleconsultation ( phone or computer consultation) followed at 6 months of a face-to-face consultation. Patients will be monitored in accordance with routine practice.
  The Teleconsultation (TC) group will be composed of patients for whom the consultation initially scheduled in the presence of the diabetologist has been replaced by a teleconsultation due to the availability of diabetologists whose activity is focused on the management of Covid-19 negative patients.
  The Face-to-Face group will be composed of patients for whom the consultation initially scheduled in the presence of the diabetologist was postponed by 6 months due to the activity of some diabetologists entirely redirected towards the management of Covid-19 positive patients.

SECONDARY OUTCOMES:
HbA1C measured at 6 months post-telemedicine consultation for the TC group / post-cancellation of the face-to-face consultation for the P group. | HbA1C will be measured at visit V2 (6 months after inclusion visit)=through study completion, an average of 6 months
Total number of patients inaccessible to teleconsultation and number of patients inaccessible by type of associated reason. | Total number of patients inaccessible to teleconsultation will be collected through study completion, an average of 6 months.
Number of complications: severe hypoglycemia, ketoacidosis, myocardial infarction, stroke, foot ulcer. | Number of complications through study completion, an average of 6 months.
Results of patient satisfaction questionnaire. | Patients will respond to the questionnaires either at the end of study (6 months after inclusion) or in the month following the teleconsultation.
  This questionnaire is not a score on a scale, there is no minimum or maximum values.
Results of doctor satisfaction questionnaire. | Physician will respond to the questionnaires at study completion, 6 months after the inclusion visit.
  This questionnaire is not a score on a scale, there is no minimum or maximum values.
Number of patients infected with Covid-19 (positive smear by RT-PCR for SARS-CoV-2 virus). | Number of patients infected with Covid-19 during the study (6 months).
Number of conventional hospitalizations, in intensive care and deaths. | Number of conventional hospitalizations, in intensive care and deaths during the study (6 months).

CONTACTS AND LOCATIONS:
Locations (1):
- Hôpitaux Universitaires de Strasbourg, Strasbourg, France

IPD SHARING:
Plan to Share IPD: No